CLINICAL TRIAL: NCT05741385
Title: Profiling Study for the Hepatic Cytochrome P450 (CYP) Isozymes CYP1A2, CYP2C9, CYP2C19, CYP2D6 and CYP3A in Healthy Subjects and in Patients With Stage 4 (F4) Liver Fibrosis / Cirrhosis by the Combined Administration of the Probe Substrates (the Cocktail) Caffeine, Warfarin, Omeprazole, Metoprolol, and Midazolam
Brief Title: A Study to Compare How Different Substances (Caffeine, Warfarin, Omeprazole, Metoprolol, and Midazolam) Are Handled by the Body of Healthy People and People With Liver Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0352-2190
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Caffeine; Warfarin; Omeprazole; Metoprolol; Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Healthy participants (Experimental): Every participant receives a cocktail of Caffeine, Warfarin sodium, Omeprazole, Metoprolol, Midazolam.
  Interventions: Drug: Caffeine; Drug: Warfarin sodium; Drug: Omeprazole; Drug: Metoprolol; Drug: Midazolam
- Group 2: F4 Child-Turcotte-Pugh class A (Child-Pugh A) participants (compensated) (Experimental): Every participant receives a cocktail of Caffeine, Warfarin sodium, Omeprazole, Metoprolol, Midazolam.
  Compensated=without any disease symptoms
  Interventions: Drug: Caffeine; Drug: Warfarin sodium; Drug: Omeprazole; Drug: Metoprolol; Drug: Midazolam
- Group 3: F4 Child-Turcotte-Pugh class B (Child-Pugh B) participants (decompensated) (Experimental): Every participant receives a cocktail of Caffeine, Warfarin sodium, Omeprazole, Metoprolol, Midazolam.
  Decompensated= with disease symptoms like aszites, variceal bleeding, hepatic encephalopathy, hepato-renal syndrome
  Interventions: Drug: Caffeine; Drug: Warfarin sodium; Drug: Omeprazole; Drug: Metoprolol; Drug: Midazolam

INTERVENTIONS:
Drug: Caffeine — Caffeine
Drug: Warfarin sodium — Warfarin sodium
Drug: Omeprazole — Omeprazole
Drug: Metoprolol — Metoprolol
Drug: Midazolam — Midazolam

SUMMARY:
This study is open to healthy adults and adults with liver cirrhosis. The purpose of this study is to compare how different medicines are handled by the body in people with and without liver cirrhosis. The study measures if the approved medicines caffeine, warfarin,omeprazole, metoprolol, and midazolam are processed differently in people with liver cirrhosis than in people without liver cirrhosis. This study will help to understand how new medicines being developed are handled by the body in people with liver cirrhosis.

There are 3 groups in this study: people without liver cirrhosis, people with mild liver cirrhosis, and people with moderate liver cirrhosis. All participants get 1 dose each of caffeine, warfarin, omeprazole, metoprolol, and midazolam by mouth. The participants with liver cirrhosis continue their regular treatment for the condition during the study.

Participants are in the study for about 1 month. During this time, they visit the study site 5 times. For 1 of the visits, participants stay overnight for 2 nights at the study site. To assess the main study endpoint, the doctors take frequent blood samples from the participants. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria

Healthy subjects and F4 liver cirrhosis patients:

* Signed and dated written informed consent in accordance with the International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Either male subject, or female subject who meets any of the following criteria for a highly effective contraception from at least 30 days before the first administration of trial medication until 30 days after trial completion:

  * Use of combined (estrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal, or transdermal), plus condom
  * Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants), plus condom
  * Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
  * Sexually abstinent
  * A vasectomised sexual partner who received medical assessment of the surgical success (documented absence of sperm) and provided that the partner is the sole sexual partner of the trial participant
  * Surgically sterilised (including hysterectomy)
  * Postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of follicle-stimulating hormone (FSH) above 40 units per liter (U/L) and estradiol below 30 nanograms per liter (ng/L) is confirmatory)
* Not taking any components in the cocktail within 4 weeks of enrolment (except from caffeine: methylxanthine-containing drinks or foods such as coffee, tea, cola, energy drinks, or chocolate are not allowed within 48 hours (h) before and during the inhouse confinement at the trial site)

Healthy subjects only:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 75 years (inclusive)
* Body mass index (BMI) of 18.5 to 35 kilograms per meter squared (kg/m2) (inclusive). A BMI of ≥ 30 is no exclusion criterion when the subject can be considered healthy apart from the elevated BMI
* further inclusion criteria apply

F4 liver cirrhosis patients only

* Male and female subjects, 18 to 75 years
* BMI of 18.5 to 40.0 kg/m2 (inclusive)
* Stable treatment for at least 4 weeks prior to taking the cocktail. Furthermore, patients can only be included into the trial a) if they are in constant specialist care at the timepoint of enrollment into the study and b) if they are willing to continue to be in specialist care after participation in the 0352.2190 study
* further inclusion criteria apply

Exclusion criteria

Healthy subjects and F4 liver cirrhosis patients:

* Subjects already taking any components in the cocktail within 4 weeks before cocktail administration (except from caffeine: methylxanthine-containing drinks or foods such as coffee, tea, cola, energy drinks, or chocolate are not allowed within 48 h before and during the in-house confinement at the trial site)
* Subjects with any other condition that would preclude administration of caffeine, warfarin, omeprazole, metoprolol, and midazolam (i.e., contraindicated as per Summary of Product Characteristics (SmPC)), such as hypersensitivity to active ingredient or any of the excipients or to any beta receptor blockers
* Repeated measurement of systolic blood pressure outside the range of 90 to 150 millimeter of mercury (mmHg), diastolic blood pressure outside the range of 50 to 95 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Relevant (other than Hepatitis B virus (HBV) or Hepatitis C virus (HCV)) chronic or acute infections (including an ongoing severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection)
* Patients receiving antiviral therapy at the time of inclusion into the trial
* further exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g., studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https:// www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study aimed to investigate whether the metabolic activity of selected CYP isozymes differs between F4 liver cirrhosis patients receiving standard therapy and healthy subjects. It was planned that 12 healthy subjects, 12 compensated F4 Child-Pugh A patients and a minimum of 6 decompensated Child-Pugh B patients following clinical confirmation enter the study. Due to insufficient enrollment only 4 patients, all from Child-Pugh A cohort, were entered into the trial.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated
Groups:
- Child-Pugh A: Patients with compensated liver cirrhosis and advanced fibrosis grade F4 and hepatic impairment that met the criteria for Child-Pugh A received a drug cocktail of caffeine, warfarin, omeprazole, metoprolol and midazolam.
  The drug cocktail was given as single oral dose of 100 mg caffeine (2 tablets), 5 mg warfarin sodium (1 tablet), 20 mg omeprazole (1 tablet), 50 mg metoprolol (1 tablet) and 2 mg/mL oral solution midazolam, with 240 mL of water after a standardized breakfast on Day 1.
Period: Overall Study
Arm/Group | Child-Pugh A
Started | 4
Completed (Completed planned observation time) | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All subjects who signed informed consent and were treated with study drug.
Arm/Group | Child-Pugh A
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.8 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Time Curve of Caffeine, Omeprazole and Metoprolol in Plasma Over the Time Interval From 0 to 24 Hours (AUC0-24)
Description: Area under the concentration time curve of caffeine, omeprazole and metoprolol in plasma over the time interval from 0 to 24 hours (AUC0-24) is reported.
Time Frame: 2 hours before drug administration and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48-72 and 96 (+/-12) hours after drug administration.
Population: Pharmacokinetic parameter analysis set (PKS): All subjects in the treated set (TS) who provide at least one PK endpoint that was defined as primary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/milliliter
Arm/Group | Child-Pugh A
Number analyzed (Participants) | 4
Hour*nanogram/milliliter
  Caffeine | 20600 (37.3)
  Omeprazole | 1520 (164)
  Metoprolol | 287 (71.1)

2. Primary Outcome: Area Under the Concentration Time Curve of Midazolam in Plasma Over the Time Interval From 0 to 24 Hours (AUC0-24)
Description: Area under the concentration time curve of midazolam in plasma over the time interval from 0 to 24 hours (AUC0-24) is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*picogram/milliliter
Arm/Group | Child-Pugh A
Number analyzed (Participants) | 4
Hour*picogram/milliliter | 31200 (51.1)

3. Primary Outcome: Area Under the Concentration Time Curve of R-warfarin and S-warfarin in Plasma Over the Time Interval From 0 to 96 Hours (AUC0-96)
Description: Area under the concentration time curve of R-warfarin and S-warfarin in plasma over the time interval from 0 to 96 hours (AUC0-96) is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/milliliter
Arm/Group | Child-Pugh A
Number analyzed (Participants) | 4
Hour*nanogram/milliliter
  R-warfarin | 11200 (18.3)
  S-warfarin | 5350 (24.7)

4. Primary Outcome: Maximum Measured Concentration of Caffeine, Omeprazole, Metoprolol, R-warfarin and S-warfarin in Plasma (Cmax)
Description: Maximum measured concentration of caffeine, omeprazole, metoprolol, R-warfarin and S-warfarin in plasma (Cmax) is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter
Arm/Group | Child-Pugh A
Number analyzed (Participants) | 4
Nanogram/milliliter
  Caffeine | 2650 (23.4)
  Omeprazole | 487 (67.9)
  Metoprolol | 73.9 (72.3)
  R-warfarin | 225 (26.3)
  S-warfarin | 226 (26.8)

5. Primary Outcome: Maximum Measured Concentration of Midazolam in Plasma (Cmax)
Description: Maximum measured concentration of midazolam in plasma (Cmax) is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram/milliliter
Arm/Group | Child-Pugh A
Number analyzed (Participants) | 4
Picogram/milliliter | 9520 (38.9)

ADVERSE EVENTS:
Time Frame: Adverse events and all-cause mortality: From administration of drug cocktail plus residual effect period, up to 9 days.
Description: Treated Set (TS): All subjects who signed informed consent and were treated with study drug.
Arm/Group | Child-Pugh A
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 2/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Child-Pugh A (N=4)
Atrioventricular block first degree (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights

DOCUMENTS (2):
  • Study Protocol (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT05741385/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT05741385/SAP_001.pdf